CLINICAL TRIAL: NCT01616199
Title: Phase 1/2 Study of PI-3K Inhibition With PX-866 Combined With Vemurafenib (BRAF Inhibitor) in Patients With BRAF-mutant Cancer Including Advanced Melanoma
Brief Title: Study of PX-866 and Vemurafenib in Patients With Advanced Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Cascadian Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PX-866-007
Record Dates: First submitted 2012-06-06; First posted 2012-06-11 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2015-07

CONDITIONS: Advanced BRAF-mutant Cancers
Keywords: PX-866; BRAF-mutant cancers; Advanced melanoma; BRAF inhibitor; Vemurafenib; Zelboraf; PI-3K inhibitor
MeSH Terms: interventions — PX-866; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1 Dose Escalation of PX-866 + vemurafenib (Experimental): PX-866 given with vemurafenib
  Interventions: Drug: PX-866; Drug: vemurafenib
- Phase 2 Combination PX-866 + vemurafenib (Experimental): PX-866 given with vemurafenib
  Interventions: Drug: PX-866; Drug: vemurafenib
- Phase 2 Single-agent vemurafenib (Active Comparator): vemurafenib given as a single agent
  Interventions: Drug: vemurafenib

INTERVENTIONS:
Drug: PX-866 — Phase 1 dose escalation: PX-866 in combination administered orally every day in 28-day cycles until progression or unacceptable toxicity.
  Phase 2 combination: PX-866 and vemurafenib administered every day in 28 day cycles until progression or unacceptable toxicity.
  Phase 2 single-agent: vemurafenib administered orally at labeled dose every day in 28 day cycles until progression or unacceptable toxicity.
  Other Names: PI-3K inhibitor
  Arms: Phase 1 Dose Escalation of PX-866 + vemurafenib; Phase 2 Combination PX-866 + vemurafenib
Drug: vemurafenib — vemurafenib is a B-Raf enzyme inhibitor
  Other Names: Zelboraf

SUMMARY:
The purpose of the phase 1 portion of the study is to determine the maximally tolerated dose (MTD) or recommended dose (RD) and the safety/tolerability of PX-866 in combination vemurafenib in patients with any advanced BRAF-mutant cancer.

The purpose of the phase 2 portion of the study is to compare progression free survival (PFS), antitumor activity (response rate), disease control rate (DCR), and the safety and tolerability of PX-866 in combination with vemurafenib vs. vemurafenib alone in patients with advanced BRAF-mutant melanoma at the doses recommended from Phase 1.

DETAILED DESCRIPTION:
This is a Phase 1 / 2 open-label study of PX-866 given in combination with vemurafenib to patients with BRAF-mutant cancer, including advanced melanoma.

Phase 1 will use a 3+3 dose escalation design to evaluate up to three dose levels of PX-866 in combination with up to two dose levels of vemurafenib in order to identify the maximal tolerated dose/recommended dose (MTD/RD) of both PX-866 and vemurafenib to be used in Phase 2. Vemurafenib will be administered orally twice per day on days 1-28 of all cycles except cycle 1, where vemurafenib will be administered on days 9-28 to allow for PK assessments). PX-866 will be administered once per day on days 1-28 of each cycle.

Phase 2 will evaluate the antitumor activity and safety of PX-866 given to patients randomized 2:1 to receive combination with vemurafenib at the doses recommended from Phase 1 compared with vemurafenib alone administered at the approved dose orally BID. All treatments will be administered on a 28-day cycle.

Patients randomized to receive single-agent vemurafenib may cross-over to receive the combination treatment at the time of progression. Patients will be evaluated for progression approximately every 8 weeks for the initial 24 weeks and every 12 weeks thereafter. All patients with stable disease (SD) or better, will receive repeat cycles until disease progression (PD), unacceptable toxicity, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years at time of consent
* If a sexually active male or a sexually active female of child-bearing potential, agrees to use a highly effective form of contraception (including birth control pills, barrier device, or intrauterine device)from the time of consent 90 days following the last dose of study drug
* If female of child-bearing potential, negative pregnancy test
* For Phase 1: must have histologically or cytologically-confirmed advanced cancer that is BRAF mutation-positive (V600E or V600K) for which there is no remaining standard therapy with curative potential. Patients must have disease sites amenable to biopsy. For Phase 2: must have histologically or cytologically-confirmed BRAF mutation-positive (V600E or V600K) advanced (defined as unresectable Stage IIIC or IV) melanoma that has not been treated with a selective BRAF inhibitor
* For Phase 1: must have measurable or non-measurable disease. For Phase 2: must have measurable disease per RECIST 1.1
* For Phase 1: no restriction on number of prior therapy regimens. For Phase 2: the following restrictions on prior therapy apply: 1) must not have been treated with a selective BRAF inhibitor and must not have had more than 2 prior treatment regimens for advanced metastatic disease; 2) must have completed prior cytotoxic chemotherapy a minimum of 4 weeks prior to starting PX-866 and/or vemurafenib (except for BCNU and/or mitomycin C, which must have been completed a minimum of 6 weeks prior to starting therapy). Prior biologic therapy and localized radiation therapy must have been completed a minimum of 2 weeks prior to starting therapy.
* All toxicities related to prior cancer therapies other than alopecia must have resolved to Grade 1 or less
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* In the opinion of the clinical investigator, life expectancy > 3 months
* Adequate hematologic function
* Adequate hepatic function
* Serum creatinine < 2.0 mg/dL
* Adequate cardiac function
* Corrected QTc must be <480 milliseconds

Exclusion Criteria:

* May not be receiving any other investigational agents
* Active central nervous system (CNS) metastases are excluded. Patients with a history of CNS metastasis, who have been treated prior to enrollment, must be stable for eight weeks after completion of treatment. These patients must have undergone appropriate imaging studies and currently be on a stable, lowest possible dose of steroids
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PX-866 or vemurafenib
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Uncorrectable electrolyte abnormalities or long QT syndrome
* Poorly controlled diabetes mellitus
* Pregnant, breastfeeding, or planning to become pregnant
* Known to be human immunodeficiency virus (HIV)-positive
* Inability to swallow pills
* Previous treatment with a phosphatidylinositol-3-kinase (PI-3K) inhibitor
* Any other significant medical or psychiatric condition that in the opinion of the investigator renders the patient inadequate for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (phase 1) | 28 days
Progression-free survival (PFS) (phase 2) | 56 days

SECONDARY OUTCOMES:
Plasma concentrations of PX-866 and metabolites (phase 1) | 44 days
Objective Response Rate (ORR)(phase 2) | 56 days
Disease Control Rate (DCR)(phase 2) | 56 Days
Plasma concentrations of vemurafenib (phase 1) | 44 days

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - New York University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee